CLINICAL TRIAL: NCT04583852
Title: A Single Center, Randomized, Double-blind and Placebo Controlled Clinical Study to Evaluate the Efficacy and Safety of Brightening Micro-needle Patch on Facial Solar Lentigines
Brief Title: Evaluate the Efficacy and Safety of Brightening Micro-needle Patch on Facial Solar Lentigines
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Panion & BF Biotech Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PBF-MN-01
Record Dates: First submitted 2020-09-10; First posted 2020-10-12 (Actual); Last update posted 2022-05-24 (Actual); Status verified 2022-05

CONDITIONS: Solar Lentigines
Keywords: Solar Lentigines; Micro-needle patch

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- brightening micro-needle patch (Experimental): apply brightening micro-needle patch to one of the two assigned spots on the face according to the instructions on the package
  Interventions: Other: AIVÍA, Ultra-Brightening Spot Micro-needle Patch
- Placebo (Placebo Comparator): apply placebo micro-needle patch to another one of the two assigned spots on the face according to the instructions on the package
  Interventions: Other: Placebo Micro-needle Patch

INTERVENTIONS:
Other: AIVÍA, Ultra-Brightening Spot Micro-needle Patch — a dissolving micro-needle patch, contains active ingredients
  Arms: brightening micro-needle patch
Other: Placebo Micro-needle Patch — matching placebo will be provided as a dissolving micro-needle patch
  Arms: Placebo

SUMMARY:
This is a single center, randomized, double-blind and placebo controlled clinical study to evaluate the efficacy and safety of brightening microneedle patch on facial solar lentigines. Subjects who are 30 to 65-year-old with solar lentigines on their faces will receive brightening microneedle patches on facial solar lentigines once a day for 4 weeks. Afterwards, facial images and skin detectors will be used to analysis their skin, according to various skin tone indexes and skin response score sheets.

DETAILED DESCRIPTION:
Method: 35 subjects, Fitzpatrick Skin Type II to IV. Each subject has at least two brown solar lentigines on the face, and the two spots are independent, each with a clear boundary and diameter ≥ 0.5 cm.

This trial includes 1 screening visit (Day -1), wash-out period (2 weeks before the trial), trial period (4 weeks in total), and 3 return visits for detecting (baseline detecting at the end of the wash-out period, the 2nd week and the 4th week of the trial period).

ELIGIBILITY:
Inclusion Criteria

1. Men or women between 30 and 65 years old (inclusive);
2. The PI determines the subject's skin type as Fitzpatrick Skin Type II to IV;
3. The PI's diagnosis is that the subject has at least two brown solar lentigines on the face, and the two spots are independent, each with a clear boundary and diameter ≥ 0.5 cm;
4. The subject can understand and follow the requirements, instructions and restriction of the plan;
5. The subject signs patient consent form in writing.

Exclusion Criteria

1. The PI's diagnosis is that the subject has tissue mutation, inflammation or other lesions on the face;
2. Those who have received aggressive facial treatments within the past six months, including laser, IPL, RF (radio frequency), HIFU(high-intensity focus ultrasound), or dermal filler injection;
3. Those with a history of chronic skin diseases or autoimmune diseases, such as atopic dermatitis, psoriasis, chronic urticaria, vitiligo, rosacea, keloid and so forth;
4. Those who have a history of allergies to the product ingredients of the brightening micro-needle patch, the moisturizer or the sunscreen provided by the trial;
5. Pregnant or lactating women;
6. Those who have used facial blemish-lightening products (such as products claiming to have whitening or blemish-lightening effects), topical or oral whitening drugs within 21 days before entering the trial;
7. Those who have smoking habits within 12 months before entering the trial;
8. Those who have used any skin medication on the face within 30 days before entering the trial, determined by the PI to have effect on this study;
9. Those who have participated in other clinical trials within 30 days before entering the trial;
10. Those who are currently undergoing medical treatment and their ability to participate in this trial will be affected;
11. Those who the PI considers to be unsuitable to join this trial.

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2020-09-14 (Actual); Primary Completion 2021-01-08 (Actual); Study Completion 2021-01-25 (Actual)

PRIMARY OUTCOMES:
the percentage change of skin tone index ITA° value of facial solar lentigines from baseline | 4 week
  measure L* (luminance) and b* (yellow/blue component) values at baseline and 4th week by color meter (CR-400 Chroma Meter) to assess the ITA° percentage change. (ITA°=tangent arc((L*-50)/b*) 180/3.14159)

SECONDARY OUTCOMES:
the value change of skin tone index ITA° value of facial solar lentigines from baseline | 4 week
  measure L* (luminance) and b* (yellow/blue component) values by color meter (CR-400 Chroma Meter) at baseline and 4th week to assess the ITA° value change. (ITA°=tangent arc((L*-50)/b*) 180/3.14159)
the value change of skin tone index ITA° value of facial solar lentigines from baseline | 2 week
  measure L* (luminance) and b* (yellow/blue component) values by color meter (CR-400 Chroma Meter) at baseline and 2nd week to assess the ITA° value change. (ITA°=tangent arc((L*-50)/b*) 180/3.14159)
the value change of melanin index of facial solar lentigines from baseline | 2 week
  measure the melanin index by CK Mexameter at baseline and 2nd week
the value change of melanin index of facial solar lentigines from baseline | 4 week
  measure the melanin index by CK Mexameter at baseline and 4th week
the percentage change of melanin index of facial solar lentigines from baseline | 2 week
  measure the melanin index by CK Mexameter at baseline and 2nd week
the percentage change of melanin index of facial solar lentigines from baseline | 4 week
  measure the melanin index by CK Mexameter at baseline and 4th week
rating the improvement of facial solar lentigines on the facial image taken by VISIA, skin analysis imaging system | 2 week
  use Physician Global Assessment (PGA) to assess the percentage improvement of lesions using VISIA images , with a scale of -1 to 5
rating the improvement of facial solar lentigines on the facial image taken by VISIA, skin analysis imaging system | 4 week
  use Physician Global Assessment (PGA) to assess the percentage improvement of lesions using VISIA images , with a scale of -1 to 5
assessing the value change of skin tone index L*a*b* of facial solar lentigines from baseline | 2 week
  determine the facial spot color index L*a*b* by color meter (CR-400 Chroma Meter) at baseline and 2nd week
assessing the value change of skin tone index L*a*b* of facial solar lentigines from baseline | 4 week
  determine the facial spot color index L*a*b* by color meter (CR-400 Chroma Meter) at baseline and 4th week
assessing the percentage change of skin tone index L*a*b* of facial solar lentigines from baseline | 2 week
  determine the facial spot color index L*a*b* by color meter (CR-400 Chroma Meter) at baseline and 2nd week
assessing the percentage change of skin tone index L*a*b* of facial solar lentigines from baseline | 4 week
  determine the facial spot color index L*a*b* by color meter (CR-400 Chroma Meter) at baseline and 4th week
assessing the patches safety on the skin by adverse reactions | through study completion, an average of 4 weeks
  assess by the incidence of adverse reactions
assessing the patches safety on the skin by subject diary | through study completion, an average of 4 weeks
  assess by subject diary
assessing the patches safety on the skin by skin response | through study completion, an average of 4 weeks
  assess by skin response score sheets
assessing the subjects' compliance with the trial by subjects' return visits | through study completion, an average of 4 weeks
  assess subjects' compliance by the number of the subjects' return visits
assessing the subjects' compliance with the trial by subject diary | through study completion, an average of 4 weeks
  assess subjects' compliance by subject diary
assessing the subjects' compliance with the trial by the number of patches packages returned | through study completion, an average of 4 weeks
  assess subjects' compliance by the number of patches packages returned by the subjects
assessing the subjects' feedback of the patches | through study completion, an average of 4 weeks
  assess the questionnaire completed by the subjects. Items in the questionnaire include satisfaction, patch usability, patch shape, patch size, skin quality after using the patch, issues with product use, etc.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Dermatology, National Taiwan University, Taipei, Taiwan